CLINICAL TRIAL: NCT02087800
Title: Effect of Smoking on Stress-Induced Allopregnanolone Response in Women by Menstrual Phase
Brief Title: Smoking, Stress & Allopregnanolone Response
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2013NTLS120
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-08

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; smoking abstinence; allopregnanolone
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- F Phase Lab session: Potential participants will complete an interview over the phone, followed by an in clinic office visit, to assess eligibility. Those who meet eligibility criteria will be invited to attend two four-hour lab sessions. Lab sessions will occur in the F (F phase lab session) and L phases (L phase lab session) of menses. In this arm, the F phase lab session will be first. Followed by the L phase lab session.
  Interventions: Behavioral: F phase lab session; Behavioral: L phase lab session
- L Phase Lab Session: Potential participants will complete an interview over the phone, followed by an in clinic office visit, to assess eligibility. Those who meet eligibility criteria will be invited to attend two four-hour lab sessions. Lab sessions will occur in the F (F phase lab session) and L phases (L phase lab session) of menses. In this arm, the L phase lab session will be first. Followed by the F phase lab session.
  Interventions: Behavioral: F phase lab session; Behavioral: L phase lab session

INTERVENTIONS:
Behavioral: F phase lab session — F phase sessions will occur three to seven days post the onset of menses. It will include blood draws, an acute stressor and completion of questionnaires.
Behavioral: L phase lab session — L phase sessions will occur six to ten days prior to the onset of the next expected menses. It will include blood draws, an acute stressor and completion of questionnaires.

SUMMARY:
This study aims to characterize the effect of smoking on stress-induced allopregnanolone (ALLO) response in women by menstrual phase. The investigators hypothesize that women who smoke will have a blunted ALLO response to stress.

DETAILED DESCRIPTION:
Cigarette smoking persists as the leading cause of preventable morbidity and mortality. Thus, finding ways to maximize quitting behavior is critical. Women have a more difficult time achieving smoking abstinence than men. The risk for smoking relapse appears to vary by menstrual phase such that the follicular phase is associated with greater risk compared to the luteal phase. Women are also more likely to smoke in response to stressful stimuli than men. Allopregnanolone (ALLO) is a stress-reducing neuroactive steroid that is primarily metabolized from the sex hormone progesterone and, therefore, varies by menstrual phase in women. Recent preclinical literature has indicated that ALLO may protect against drug abuse behaviors. Unfortunately, ALLO remains largely unexplored in clinical samples containing women.

In this study we aim to characterize the effect of smoking on stress-induced ALLO response in women by menstrual phase. To achieve this goal, we will recruit a sample of premenopausal women who smoke (n=30) and do not smoke (n=30) to participate in a controlled cross-over study. All participants will complete two four-hour lab sessions timed to occur in the Follicular (F; low ALLO) and Luteal (L; high ALLO) menstrual phases. Each lab session will contain an acute stressor along with a timed series of assessments including blood samples (for ALLO measurement) and self-report of mood and perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* Female between the ages of 18-40 years old
* Stable physical/mental health,
* Self-report of regular menstrual cycles,
* Self-report of either smoking either current or never smoking,
* English fluency,
* Ability to provide informed consent

Exclusion Criteria:

* Self-report of current use of illicit drugs, other tobacco products, nicotine, or smoking cessation medications,
* Current or recent pregnancy or breastfeeding,
* Current or recent use of exogenous hormones (including birth control pills),
* Current or recent use of psychotropic medications.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between the ages of 18 and 40 who either smoke or do not smoke.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in allopregnanolone levels | 6 weeks
  The change in ALLO after delivery of the acute stressor will be analyzed.

SECONDARY OUTCOMES:
Change in mood | 6 weeks
  We will analyze ALLO levels and mood to see if there is an association between the two.
Change in stress level | 6 weeks
  We will analyze ALLO levels and perceived stress level to see if there is an association and whether stress changes as ALLO levels change.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Allen, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Tobacco Research Program, Minneapolis, Minnesota, United States